CLINICAL TRIAL: NCT03715387
Title: Malar Bags After Lower Lid Blepharoplasty and Facelift: A Randomized Controlled Trial of the Effects of Tacrolimus
Brief Title: Tacrolimus for Malar Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Richard Warren, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: H17-02969
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Edema Face
MeSH Terms: interventions — Tacrolimus; Ointments; polysporin ointment; bacitracin, polymyxin B drug combination

STUDY DESIGN:
Intervention Model Description: Patients will serve as their own self matched controls with one study cheek and one control cheek.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will receive a container for each cheek where the contents will be randomized between the study ointment and the control ointment. Only one investigator will have knowledge of the contents. The care providor, patient, and assessor will all be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus Treatment (Experimental): Tacrolimus Topical 0.1% Topical Ointment
  Interventions: Drug: Tacrolimus Topical 0.1% Topical Ointment
- Control (Placebo Comparator): Patients will be self matched controls with one cheek receiving the study ointment and the other receiving a control ointment (polysporin ointment).
  Interventions: Drug: Polysporin Ointment

INTERVENTIONS:
Drug: Tacrolimus Topical 0.1% Topical Ointment — Topical tacrolimus ointment
  Other Names: Protopic
  Arms: Tacrolimus Treatment
Drug: Polysporin Ointment — Polysporin ointment
  Other Names: Polysporin
  Arms: Control

SUMMARY:
Elective lower eyelid surgery is a common cosmetic procedure. Facial swelling is a common complication. Studies suggest that this facial swelling is part of a complex inflammatory process. Topical tacrolimus has long been used to treat various inflammatory skin disorders. By combining our knowledge of facial swelling and tacrolimus mechanism of action, we can hypothesize that it can be used as a treatment to prevent this post-operative swelling. The purpose of this project is to apply topical tacrolimus to one of the patient's cheeks following facial surgery and compare the incidence of facial swelling to the opposite side control cheek.

DETAILED DESCRIPTION:
1.0 Purpose:

To perform a randomized controlled trial to determine if topical tacrolimus ointment reduces incidence or severity of post-operative facial edema and malar bags after elective blepharoplasty and/or facelift.

2.0 Hypothesis:

Topical tacrolimus will reduce the incidence and severity of post-operative facial edema presenting as malar bags after blepharoplasty and/or facelift.

3.0 Justification:

Elective blepharoplasty is the fourth most common cosmetic procedures performed in North America. According to a report published by the American Society of Plastic Surgery, eye lid surgery accounted for 209,000 out of the 1.7 million cosmetic surgical procedures performed in 2016. Additionally, the number of eye lid surgeries rose 2% in 2016 compared to 2015 [ref 1].

Recurrent or worsened malar bags is a common complication of lower lid surgery. Studies suggest that post-operative lymphedema is a possible cause of these malar bags. Recent research into lymphedema pathophysiology shows that post-operative lymphedema is not simply a result of direct lymphatic injury, but rather a complex fibroproliferative inflammatory process.

Topical tacrolimus has long been used to treat various inflammatory skin disorders such as atopic dermatitis and psoriasis safely and effectively. By combining our knowledge of lymphedema pathophysiology and tacrolimus mechanism of action, we can hypothesize that it can be effectively used as a treatment to prevent post-operative malar bags as a result of lymphedema.

4.0 Objectives:

4.1. To apply topical tacrolimus ointment to a randomized cheek in sequential patients undergoing lower lid blepharoplasty, facelift or both and compare to the contralateral control cheek.

4.2. To determine if topical tacrolimus affects the incidence and severity of post-operative malar edema compared to the self-matched contralateral control cheek.

5.0 Research Design:

This is a double blinded randomized controlled trial involving an initial surgery followed by random topical drug treatment that is self matched to a contralateral control side. There will be 3 follow up visits for analysis.

6.0 Statistical Analysis:

6.1 Statistical Considerations

The primary endpoint is post operative malar edema which typically occurs 10-20% of the time following lower lid blepharoplasty and/or facelift procedures. If we expect to reduce the occurrence to 1-5% the number of patients required to achieve a significant result (α = 0.05 (2-sided), β = 0.20) is 40-100.

No increase in sample size has been made to account for losses to follow-up. In our practice over the past 10 years we have found that less than 1% of patients do not return for a follow-up visit.

6.2 Outcome Measures

A custom four point scale will be used to record the outcomes for each cheek:

I: No post operative edema. II: Mild post operative edema. III: Moderate post operative edema. IV: Severe post operative edema.

Example photographs will be provided to the blinded rater for each category.

6.3 Data Collection

Outcome measurements will be performed by a single observer who will be blinded to the contents of the containers and which cheek either was applied to. Data will be collected on study specific data collection forms.

7.0 Procedure

7.1 Surgical Procedure

The lower lid blepharoplasty and facelift procedures will be performed by Dr. Richard Warren in the usual fashion based on the patient's presenting problem. Specific differences in technique such as skin only excision vs fat transposition and ORL (Orbicularis Retaining Legament) division will be recorded and analyzed separately.

7.2 Tacrolimus Application

Patients will be given two containers labelled with "Right" and "Left" to be applied to their right and left cheeks respectively. The patients will apply the ointment once daily for 4 weeks post operatively. The contents of the containers will be randomized to either the treatment tacrolimus ointment or the control ointment which will be matched in colour and consistency to the tacrolimus ointment. They will be given instructions on applying the ointments based on FDA recommendations.

7.3 Choice of Tacrolimus Dose

The treatment containers will contain 0.1% tacrolimus ointment (marketed as PROTOPIC) based on FDA recommendations for adult patients. This dose of the drug is known to be sufficiently absorbed by inflamed skin reaching peak concentrations of 0.05-0.25ng/ml 3-6 hours after application. This is significantly lower than the accepted safe level of 5-20ng/ml established based on transplant research. [ref 16,17]

7.4 Post-operative Treatment

Patients will be followed post operatively in the office at 1 week, 4 weeks, and 6 months. Degree of post operative malar edema will be assessed by a single blinded observer. This will be recorded using a four point scale. Any side effects or adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral lower lid blepharoplasty, facelift, or both.
* Patients over 18 years of age.

Exclusion Criteria:

* -Patients presenting for revision surgery.
* Patients with a known allergy to tacrolimus.
* Patients taking medications that alter tacrolimus metabolism:
* Anticonvulsants: carbamazepine, phenobarbital, phenytoin
* Antibiotics: rifampicin, rifabutin
* Antifungal: clotrimazole, ketoconazole, fluconazole, itraconazole
* Ca++ channel blockers: diltiazem, nifedipine, nicardipine, verapamil
* Macrolides: erythromycin, clarithromycin, troleandomycin
* Miscellaneous: cyclosporin A, danazol, bromocriptine, cimetidine, methylprednisolone, protease inhibitors
* Patients with previously diagnosed reduced kidney function.
* Immunocompromised patients.
* Patients with a history of cutaneous facial malignancies.
* Patients with active cutaneous facial infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Malar edema | 6 months
  Development of malar edema post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Richard Warren, MD, Principal Investigator — University of British Columbia; Stahs Pripotnev, MD, Study Chair — University of British Columbia
Locations (1):
- Vancouver Plastic Surgery Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pessa JE, Garza JR. The malar septum: the anatomic basis of malar mounds and malar edema. Aesthet Surg J. 1997 Jan-Feb;17(1):11-7. doi: 10.1016/s1090-820x(97)70001-3. PMID 19327681
- [Background] Nagi KS, Carlson JA, Wladis EJ. Histologic assessment of dermatochalasis: elastolysis and lymphostasis are fundamental and interrelated findings. Ophthalmology. 2011 Jun;118(6):1205-10. doi: 10.1016/j.ophtha.2010.10.013. Epub 2011 Jan 6. PMID 21211847
- [Background] Nijhawan N, Marriott C, Harvey JT. Lymphatic drainage patterns of the human eyelid: assessed by lymphoscintigraphy. Ophthalmic Plast Reconstr Surg. 2010 Jul-Aug;26(4):281-5. doi: 10.1097/IOP.0b013e3181c32e57. PMID 20551850
- [Background] Kpodzo DS, Nahai F, McCord CD. Malar mounds and festoons: review of current management. Aesthet Surg J. 2014 Feb;34(2):235-48. doi: 10.1177/1090820X13517897. Epub 2014 Jan 15. PMID 24431347
- [Background] Cemal Y, Pusic A, Mehrara BJ. Preventative measures for lymphedema: separating fact from fiction. J Am Coll Surg. 2011 Oct;213(4):543-51. doi: 10.1016/j.jamcollsurg.2011.07.001. Epub 2011 Jul 28. No abstract available. PMID 21802319
- [Background] Ghanta S, Cuzzone DA, Torrisi JS, Albano NJ, Joseph WJ, Savetsky IL, Gardenier JC, Chang D, Zampell JC, Mehrara BJ. Regulation of inflammation and fibrosis by macrophages in lymphedema. Am J Physiol Heart Circ Physiol. 2015 May 1;308(9):H1065-77. doi: 10.1152/ajpheart.00598.2014. Epub 2015 Feb 27. PMID 25724493
- [Background] Avraham T, Zampell JC, Yan A, Elhadad S, Weitman ES, Rockson SG, Bromberg J, Mehrara BJ. Th2 differentiation is necessary for soft tissue fibrosis and lymphatic dysfunction resulting from lymphedema. FASEB J. 2013 Mar;27(3):1114-26. doi: 10.1096/fj.12-222695. Epub 2012 Nov 27. PMID 23193171
- [Background] Clavin NW, Avraham T, Fernandez J, Daluvoy SV, Soares MA, Chaudhry A, Mehrara BJ. TGF-beta1 is a negative regulator of lymphatic regeneration during wound repair. Am J Physiol Heart Circ Physiol. 2008 Nov;295(5):H2113-27. doi: 10.1152/ajpheart.00879.2008. Epub 2008 Oct 10. PMID 18849330
- [Background] Zampell JC, Yan A, Elhadad S, Avraham T, Weitman E, Mehrara BJ. CD4(+) cells regulate fibrosis and lymphangiogenesis in response to lymphatic fluid stasis. PLoS One. 2012;7(11):e49940. doi: 10.1371/journal.pone.0049940. Epub 2012 Nov 20. PMID 23185491
- [Background] Zhang B, Wang J, Gao J, Guo Y, Chen X, Wang B, Gao J, Rao Z, Chen Z. Alternatively activated RAW264.7 macrophages enhance tumor lymphangiogenesis in mouse lung adenocarcinoma. J Cell Biochem. 2009 May 1;107(1):134-43. doi: 10.1002/jcb.22110. PMID 19241443
- [Background] Sehgal VN, Srivastava G, Dogra S. Tacrolimus in dermatology-pharmacokinetics, mechanism of action, drug interactions, dosages, and side effects: part I. Skinmed. 2008 Jan-Feb;7(1):27-30. doi: 10.1111/j.1540-9740.2007.06485.x. PMID 18174798
- [Background] Gardenier JC, Kataru RP, Hespe GE, Savetsky IL, Torrisi JS, Nores GD, Jowhar DK, Nitti MD, Schofield RC, Carlow DC, Mehrara BJ. Topical tacrolimus for the treatment of secondary lymphedema. Nat Commun. 2017 Feb 10;8:14345. doi: 10.1038/ncomms14345. PMID 28186091